CLINICAL TRIAL: NCT02767024
Title: Intravenous Vasodilator vs. Inotropic Therapy in Patients With Heart Failure Reduced Ejection Fraction and Acute Decompensation With Low Cardiac Output: A Single Center, Randomized, Non-Blinded, and Parallel Study (PRIORITY-ADHF Study)
Brief Title: Intravenous Vasodilator vs. Inotropic Therapy in Patients With Heart Failure
Acronym: PRIORITY-ADHF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Mario Garcia, Professor, Cardiology, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-3586
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Nitroprusside; Dobutamine; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium Nitroprusside (Experimental): Dose titration will start at 25 μg/min and increased by 25 μg every 5 minutes to maximal dose of 400 μg/min while maintaining SBP ≥ 90 mmHg. Every 5 minutes, the Pulmonary Capillary Wedge Pressure (PCWP), SBP will be measured. If PCWP > 16 mmHg while maintaining SBP ≥ 90 mmHg, the investigator will proceed to titrate dose with the goal to achieve the target of PCWP ≤ 16 mmHg and Cardiac Index (CI) > 2.2 L·min-1·m-2, or maximal infusion dose has been reached, whichever comes earliest. Continuous intravenous furosemide infusion dose will be maintained by protocol.
  Interventions: Drug: Sodium nitroprusside; Drug: Furosemide
- Dobutamine (Active Comparator): Dose titration will start at 2.5 μg/kg/min and increased to doses of 5, 7.5 and 10 μg/kg/min (maximal dose). Every 30 minutes, the investigator will collect Pulmonary Artery (PA) blood samples for PA sat measurement to calculate Cardiac Output (CO) and CI by Fick. If CI ≤ 2.2 L·min-1·m-2, the investigator will proceed to titrate dose until CI > 2.2 L·min-1·m-2 or maximal infusion dose has been reached, whichever comes earliest. Continuous intravenous furosemide infusion dose will be maintained by protocol.
  Interventions: Drug: Dobutamine; Drug: Furosemide

INTERVENTIONS:
Drug: Sodium nitroprusside — Sodium nitroprusside is a medication used to lower blood pressure.
  Other Names: Generic name for nitropress
  Arms: Sodium Nitroprusside
Drug: Dobutamine — Dobutamine is a direct-acting inotropic agent whose primary activity results from stimulation of the ÃŸ receptors of the heart while producing comparatively mild chronotropic, hypertensive, arrhythmogenic, and vasodilative effects.
  Arms: Dobutamine
Drug: Furosemide — Furosemide is a prescription drug used to treat hypertension (high blood pressure) and edema. Learn about side effects, warnings, dosage, and more.
  Other Names: Generic name for Lasix

SUMMARY:
Single center, prospective, randomized, non-blinded research study comparing intravenous vasodilator infusion vs. inotropic infusion in patients admitted to the hospital or in the emergency room at Montefiore Medical Center presenting with the diagnosis of acute decompensated systolic heart failure with low cardiac output but no hypotensive.

DETAILED DESCRIPTION:
The objective of the study is determine if the administration of diuretics with intravenous sodium nitroprusside (vasodilator therapy) in comparison to intravenous dobutamine (inotropic therapy) will lead to a reduction in the primary and secondary endpoints in patients with acute decompensated systolic heart failure with low cardiac output and no hypotensive.

ELIGIBILITY:
Inclusion Criteria:

* History of heart failure reduced ejection fraction (HFrEF), New York Heart Association (NYHA) class IV and known left ventricular ejection fraction (LVEF ) ≤ 40% within the last 6 months by any of the following imaging techniques: echocardiogram, radio-nuclear stress test, ventriculogram or cardiac magnetic resonance imaging (CMR) performed within 6 months.
* Hospitalized or presented to the emergency department for acute decompensated heart failure (ADHF) with the anticipated requirement if intravenous (IV) therapy (including IV diuretics). ADHF is defined as including all of the following measured at any time between the presentation (including the emergency department) and the end of the screening:

  1. Persistent dyspnea or orthopnea or edema at screening and at the time or randomization, despite standard background therapy for heart failure.
  2. Pulmonary congestion on chest radiograph.
  3. N-terminal pro b-type natriuretic peptide (NT-proBNP) ≥ 2000 pg/ml; for patients ≥ 75 years old or with current atrial fibrillation, NT-proBNP ≥ 3000 pg/ml.
* Clinical suspicious of low cardiac output state; consider by the presence of any of the following signs or symptoms of hypoperfusion: narrow pulse pressure, cold extremities, mental obtundation, declining renal function, and/or low serum sodium.
* Systolic blood pressure (SBP) measured ≥ 90 but < 120 mmHg at the start and the end of the screening, without use of an intravenous vasopressor therapy.
* Hemodynamic criteria: CI ≤ 2.2 L·min-1·m-2 based on CO calculated by Fick formula and PCWP ≥ 20 mmHg measured by right heart catheterization at the time of the enrollment and confirmed by Swan-Ganz measurement upon arrival to the Cardiac Care Unit (CCU).
* Able to be randomized within the first 24 hours from the presentation to the hospital, including the emergency department.

Exclusion Criteria:

* Clinical evidence of acute coronary syndrome (ACS) currently or within 30 days prior to enrollment. (Note that the diagnosis of ACS is a clinical diagnosis and that the sole presence of elevated troponin concentrations is not sufficient for a diagnosis of ACS).
* Significant, uncorrected left ventricular outflow track obstruction, such us obstructive cardiomyopathy or severe aortic stenosis (i.e. aortic valve area < 1.0 cm2 or mean gradient > 40 mmHg on prior or current echocardiogram).
* Severe mitral stenosis.
* Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated.
* Documented, prior to or at the time of the randomization, restrictive amyloid myocardiopathy or acute myocarditis or hypertrophic obstructive, restrictive or constrictive cardiomyopathy (does not include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function).
* Complex congenital heart disease.
* Significant arrhythmias, which include any of the following: sustained ventricular tachycardia; atrial fibrillation or atrial flutter with sustained heart rate > 130 beats per minute.
* Bradycardia with sustained ventricular rate < 45 beats per minute.
* Temperature > 38.5°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment.
* History of malignancy (other than localized basal cell carcinoma of the skin), treated or untreated or any terminal illness (other than heart failure) with a current life expectancy less than a year.
* Major surgery or major neurologic event including cerebrovascular events, within 30 days prior to enrollment.
* Need for mechanical circulatory support (MCS), including intra-aortic balloon pump, Extracorporeal Membrane Oxygenation (ECMO) or any ventricular assist device.
* Need for mechanical ventilatory support (endotracheal intubation or mechanical ventilation).
* Patient with chronic heart failure and inotropic-depended.
* Current (within 2 hours prior to screening) treatment with any IV vasoactive therapies, including vasodilators, inotropic agents and vasopressors.
* Patients with severe renal impairment defined as pre-randomization estimated Glomerular Filtration Rate (eGFR) < 25 ml/min/1.73m2 calculated using the simplified Modification of Diet in Renal Disease (sMDRD) equalization and/or those receiving current or planned dialysis or ultrafiltration.
* Patients with acute kidney injury defined as an increase in serum creatinine 3 times of baseline, or reduction in urine output to <0.3 mL/kg per hour for ≥12 hours, or anuria for ≥12 hours, or patients undergoing renal replacement therapy.
* Patients with Child C cirrhosis or history of cirrhosis with evidence of portal hypertension such as varices.
* Patients with acute liver failure and serum transaminase: aspartate transaminase (AST) and/or alanine transaminase (ALT) > 3 times above the upper limit of normal.
* Any major solid organ transplant recipient or planned/anticipated organ transplant within 1 year.
* Patients with hematocrit < 25%, or a history of blood transfusion within 14 days prior to screening, or active life-threatening gastrointestinal bleeding.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test. .
* History of hypersensitive to dobutamine or sodium nitroprusside.
* Inability to follow instructions or comply with follow-up procedures.
* Any other medical condition (s) that the investigator deems unsuitable for the study, including drug or alcohol use or psychiatric, behavioral or cognitive disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Arrhythmia incidence | within 72 hours after the initiation of the drug
  defined by the presence of ventricular arrhythmia (either ventricular tachycardia or ventricular fibrillation) or supraventricular arrhythmias (either recurrent or new onset of atrial fibrillation, atrial flutter or supraventricular tachycardia) with sustained heart rate ≥ 130 beats per minute
Serum troponin T release | within 72 hours after the initiation of the drug
  defined as measured serum cardiac troponin T (cTnT) with a value > 0.10 ng/ml
Hypotension incidence | within 72 hours after the initiation of the drug
  defined as ≥ 2 consecutive blood pressure measurement with SBP < 90 mmHg

SECONDARY OUTCOMES:
≥2 point improvement in the 5 point Likert dyspnea scale | within 72 hours after the initiation of the drug involved in the study
≥ 30% improvement in the 100 point global patient assessment scale | within 72 hours after the initiation of the drug involved in the study
Reduction in the Cardiac Care Unit length of stay | Up to 30 days
  Length of stay (in hours) will be defined as the index discharge date and time minus the initiation of study drug date and time.
Reduction in the hospitalization length of stay | Up to 30 days
  Length of stay (in hours) will be defined as the index discharge date and time minus the initiation of study drug date and time.
Assessment of difference in restrictive filling pattern by echocardiogram | from initiation of the of the drug involved in the study up to 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Background] Gheorghiade M, Zannad F, Sopko G, Klein L, Pina IL, Konstam MA, Massie BM, Roland E, Targum S, Collins SP, Filippatos G, Tavazzi L; International Working Group on Acute Heart Failure Syndromes. Acute heart failure syndromes: current state and framework for future research. Circulation. 2005 Dec 20;112(25):3958-68. doi: 10.1161/CIRCULATIONAHA.105.590091. No abstract available. PMID 16365214
- [Background] Heart Failure Society of America; Lindenfeld J, Albert NM, Boehmer JP, Collins SP, Ezekowitz JA, Givertz MM, Katz SD, Klapholz M, Moser DK, Rogers JG, Starling RC, Stevenson WG, Tang WH, Teerlink JR, Walsh MN. HFSA 2010 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2010 Jun;16(6):e1-194. doi: 10.1016/j.cardfail.2010.04.004. PMID 20610207
- [Background] Mebazaa A, Nieminen MS, Packer M, Cohen-Solal A, Kleber FX, Pocock SJ, Thakkar R, Padley RJ, Poder P, Kivikko M; SURVIVE Investigators. Levosimendan vs dobutamine for patients with acute decompensated heart failure: the SURVIVE Randomized Trial. JAMA. 2007 May 2;297(17):1883-91. doi: 10.1001/jama.297.17.1883. PMID 17473298
- [Background] Gage J, Rutman H, Lucido D, LeJemtel TH. Additive effects of dobutamine and amrinone on myocardial contractility and ventricular performance in patients with severe heart failure. Circulation. 1986 Aug;74(2):367-73. doi: 10.1161/01.cir.74.2.367. PMID 3731427
- [Background] Mager G, Klocke RK, Kux A, Hopp HW, Hilger HH. Phosphodiesterase III inhibition or adrenoreceptor stimulation: milrinone as an alternative to dobutamine in the treatment of severe heart failure. Am Heart J. 1991 Jun;121(6 Pt 2):1974-83. doi: 10.1016/0002-8703(91)90834-5. PMID 1852090
- [Background] Cuffe MS, Califf RM, Adams KF Jr, Benza R, Bourge R, Colucci WS, Massie BM, O'Connor CM, Pina I, Quigg R, Silver MA, Gheorghiade M; Outcomes of a Prospective Trial of Intravenous Milrinone for Exacerbations of Chronic Heart Failure (OPTIME-CHF) Investigators. Short-term intravenous milrinone for acute exacerbation of chronic heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1541-7. doi: 10.1001/jama.287.12.1541. PMID 11911756
- [Background] Abraham WT, Adams KF, Fonarow GC, Costanzo MR, Berkowitz RL, LeJemtel TH, Cheng ML, Wynne J; ADHERE Scientific Advisory Committee and Investigators; ADHERE Study Group. In-hospital mortality in patients with acute decompensated heart failure requiring intravenous vasoactive medications: an analysis from the Acute Decompensated Heart Failure National Registry (ADHERE). J Am Coll Cardiol. 2005 Jul 5;46(1):57-64. doi: 10.1016/j.jacc.2005.03.051. PMID 15992636
- [Background] Elkayam U, Tasissa G, Binanay C, Stevenson LW, Gheorghiade M, Warnica JW, Young JB, Rayburn BK, Rogers JG, DeMarco T, Leier CV. Use and impact of inotropes and vasodilator therapy in hospitalized patients with severe heart failure. Am Heart J. 2007 Jan;153(1):98-104. doi: 10.1016/j.ahj.2006.09.005. PMID 17174645
- [Background] Grant S, Aitchison T, Henderson E, Christie J, Zare S, McMurray J, Dargie H. A comparison of the reproducibility and the sensitivity to change of visual analogue scales, Borg scales, and Likert scales in normal subjects during submaximal exercise. Chest. 1999 Nov;116(5):1208-17. doi: 10.1378/chest.116.5.1208. PMID 10559077
- [Background] Allen LA, Metra M, Milo-Cotter O, Filippatos G, Reisin LH, Bensimhon DR, Gronda EG, Colombo P, Felker GM, Cas LD, Kremastinos DT, O'Connor CM, Cotter G, Davison BA, Dittrich HC, Velazquez EJ. Improvements in signs and symptoms during hospitalization for acute heart failure follow different patterns and depend on the measurement scales used: an international, prospective registry to evaluate the evolution of measures of disease severity in acute heart failure (MEASURE-AHF). J Card Fail. 2008 Nov;14(9):777-84. doi: 10.1016/j.cardfail.2008.07.188. Epub 2008 Aug 15. PMID 18995183
- [Background] Binanay C, Califf RM, Hasselblad V, O'Connor CM, Shah MR, Sopko G, Stevenson LW, Francis GS, Leier CV, Miller LW; ESCAPE Investigators and ESCAPE Study Coordinators. Evaluation study of congestive heart failure and pulmonary artery catheterization effectiveness: the ESCAPE trial. JAMA. 2005 Oct 5;294(13):1625-33. doi: 10.1001/jama.294.13.1625. PMID 16204662
- [Background] Mullens W, Abrahams Z, Francis GS, Skouri HN, Starling RC, Young JB, Taylor DO, Tang WH. Sodium nitroprusside for advanced low-output heart failure. J Am Coll Cardiol. 2008 Jul 15;52(3):200-7. doi: 10.1016/j.jacc.2008.02.083. PMID 18617068